CLINICAL TRIAL: NCT06517563
Title: An Open-Label Study to Assess the Effects of VMX-C001 in Combination With an Oral FXa DOAC on the Efficacy of Unfractionated Heparin and of VMX-C001 Alone on the Efficacy of Low Molecular Weight Heparin in Healthy Subjects
Brief Title: Effects of VMX-C001 on the Anticoagulant Effect of Different Forms of Heparin
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VarmX B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMX-C001-02; 2022-003675-41 (EudraCT Number)
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Coagulation Disorder
Keywords: Direct oral anticoagulant (DOAC); Human coagulation factor X
MeSH Terms: conditions — Hemostatic Disorders | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UFH Cohort (Experimental): Subjects will be administered 2 single doses of 5000 IU UFH i.v. on Day 1 and Day 5, oral doses of the DOAC Rivaroxaban QD from Day 2 until the morning of Day 5, and one single dose of 170 mg VMX-C001 i.v. on Day 5.
  Interventions: Drug: VMX-C001; Drug: Rivaroxaban; Drug: UFH
- LMWH Cohort (Experimental): Subjects will be administered 2 single doses of 40 mg Enoxaparin s.c. on Day 1 and Day 4, and one single dose of 170 mg VMX-C001 i.v. on Day 4.
  Interventions: Drug: VMX-C001; Drug: Enoxaparin

INTERVENTIONS:
Drug: VMX-C001 — VMX-C001 is human factor X engineered to be insensitive to factor Xa DOACs
Drug: Rivaroxaban — FXa Inhibitor
  Arms: UFH Cohort
Drug: UFH — Unfractionated Heparin
  Arms: UFH Cohort
Drug: Enoxaparin — Low Molecular Weight Heparin
  Arms: LMWH Cohort

SUMMARY:
A single centre, open-label study to assess the effects of VMX-C001 in combination with an oral FXa DOAC on the efficacy of Unfractionated Heparin (UFH) and of VMX-C001 alone on the efficacy of Low Molecular Weight Heparin (LMWH) in healthy subjects conducted in two parts:

UFH cohort: Subjects will be administered 2 single doses of 5000 IU UFH i.v. on Day 1 and Day 5, oral doses of the DOAC Rivaroxaban once daily from Day 2 until the morning of Day 5, and one single dose of 170 mg VMX-C001 i.v. on Day 5.

LMWH cohort: Subjects will be administered 2 single doses of 40 mg Enoxaparin s.c. on Day 1 and Day 4, and one single dose of 170 mg VMX-C001 i.v. on Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of any ethnic origin aged between 18 and 49 years of age, inclusive, at the time of Screening.
2. Male subjects must be willing to use appropriate contraception, such as a condom, and to refrain from sperm donation during the main study and until 90 days after study drug administration.
3. Women of child-bearing potential must agree not to attempt to become pregnant and to use a highly effective form of birth control during the main study and for 90 days after study drug administration when their sexual partner has not been vasectomized. Highly effective forms of birth control entail the use of combined (estrogen- and progestogen-containing) or progestogen-only hormonal contraception associated with inhibition of ovulation, an intrauterine device (IUD), an intrauterine hormone-releasing system (IUS) or abstinence.
4. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with documented follicle stimulating hormone [FSH] >33.4 IU/L).
5. Surgically sterile women are defined as those who have had a surgical bilateral oophorectomy with or without hysterectomy, total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, the reproductive status of the woman has to be confirmed by follow-up hormone level assessment. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
6. Subject must weigh between 60 and 120 kg, inclusive, and must have a BMI between 18.0 and 30.0 kg/m2, inclusive, at Screening and on Day -1.
7. Subject must be in good health, as determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations (congenital non hemolytic hyperbilirubinemia is acceptable).
8. Subject is willing and able to give their written informed consent to participate in the study and to abide by the study restrictions.
9. Subject has good upper limb venous access.

Exclusion Criteria:

1. The subject has taken tenoxicam in the 35 days prior to Day 1 or has taken piroxicam in the two weeks prior to Day 1.
2. The subject is receiving or requires, for any cause, any anticoagulant or antiplatelet therapy including warfarin, clopidogrel or aspirin or any other anticoagulant or antiplatelet agent or has used these therapies in the 4 weeks prior to Day 1.
3. The subject has taken any non-aspirin, non-tenoxicam, non-piroxicam non-steroidal antiinflammatory drug (NSAID) in the week prior to Day 1.
4. The subject requires or has taken during the 4 weeks prior to Day 1, vitamin K for therapeutic reasons. Vitamin K not taken for therapeutic purposes is acceptable, e.g. as part of a multivitamin supplement.
5. The subject has received any prescribed oral, systemic or topical medication, including any vaccinations, within 14 days before Day 1 (with the exception of contraceptives), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
6. The subject has used any non-prescribed systemic or topical medication (including herbal remedies) within 4 days prior to Day 1 (with the exception of oral vitamin/mineral supplements [including those that contain vitamin K when not taken for therapeutic purposes] and paracetamol), unless in the opinion of the Principal Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
7. The subject has been administered an investigational drug (new chemical or biological entity) within 4 weeks prior to Day 1 for small molecules or within 12 weeks or 5 halflives, whichever is longer, prior to Day 1 for all other types of investigational drug.
8. The subject has donated ≥500 mL blood, plasma or platelets in the 12 weeks prior to Screening or the subject has donated any blood amount within 30 days prior to Screening.
9. Because of an increased risk of thrombosis, subjects with known diabetes mellitus or a fasted glucose ≥7.0 mmol/l at Screening.
10. The subject has any bleeding diathesis, any increased risk of bleeding or, in the opinion of the Principal Investigator, is at increased risk of the consequences of bleeding including but not limited to the following:

    1. gastro-intestinal ulceration within the last 12 weeks;
    2. known or suspected oesophageal varices;
    3. vascular aneurysms or known arteriovenous malformations;
    4. history of known major intraspinal or intracerebral vascular abnormalities;
    5. history of brain, spinal or ophthalmic surgery within the last year;
    6. any intracranial hemorrhage;
    7. uncontrolled severe hypertension.
11. The subject has, in the opinion of the Principal Investigator, any increased risk of thrombosis or thromboembolism including any known thrombophilia, such as antiphospholipid syndrome, or any past history of provoked or unprovoked arterial or venous thrombosis, including thromboembolism.
12. The subject has a significant history of drug allergy, as determined by the Principal Investigator.
13. The subject has, at Screening or on Day -1, a supine blood pressure or supine pulse rate ≥ 150/95 mmHg and >100 beats per minute (bpm), respectively, or < 90/40 mmHg and 40 bpm, respectively, confirmed by a repeat assessment.
14. The subject consumes > 21 alcoholic drinks/week for men or > 14 alcoholic drinks/week for women (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1 measure [25 mL] of spirits), or has a significant history of alcoholism or drug/chemical abuse, as determined by the Principal Investigator.
15. The subject has a positive drug screen, alcohol test or cotinine test result at Screening or on Day -1, confirmed by repeat testing.
16. The female subject has a positive pregnancy test at Screening or on Day -1, or is lactating.
17. The subject currently smokes or uses nicotine-containing products. Former smokers will be eligible, provided they have not smoked for at least 4 weeks prior to administration of the study drug.
18. The subject has, or has a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological or other major disorders, as determined by the Principal Investigator.
19. The subject has a positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody test result at Screening.
20. The subject has an abnormality in the 12-lead ECG at Screening or on Day -1 that, in the judgement of the Principal Investigator may, during the main study, interfere with the interpretation of 12-lead ECG results, including average QTcF interval >450 msec for men or >470 msec for women, 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as average PR<110 msec, confirmed by a triplicate repeat ECG.
21. The subject has any other condition that, in the opinion of the Principal Investigator, would compromise the safety of the subject or the subject's ability to comply with the protocol and complete the study.
22. The subject has renal insufficiency (serum creatinine level > 1.25 times upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) of <60 mL/minute*1.73m2 at Screening or on Day -1. One re-test is allowed).
23. The subject has active liver disease (alanine transaminase [ALT]/ aspartate transaminase [AST] >1.5x ULN, or total bilirubin > 1.5x ULN at Screening or on Day -1. One re-test is allowed).
24. The subject has previously participated in a clinical study with VMX-C001.
25. The subject has any contra-indication to treatment with heparin (LMWH or UFH).

    Additional exclusion criteria for UFH Cohort only:
26. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received medication that is an inhibitor of P-glycoprotein or CYP3A4. (eg clarithromycin, erythromycin and azole-antimycotics such as ketoconazole, itraconazole, voriconazole and posaconazole or HIV protease inhibitors.) within 30 days prior to Day 1.
27. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received treatment with CYP3A4 inducers (eg St. John's wort, rifampicin, phenytoin, carbamazepine, phenobarbital within 30 days prior to Day 1.
28. Because of an effect on FXa DOACs, subjects are to be excluded if he/she receives or has received treatment with selective serotonin reuptake inhibitors (SSRIs) or selective noradrenaline reuptake inhibitors (SNRIs) within 30 days prior to Day 1.
29. The subject has any contra-indication to treatment with DOACs.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in thrombin time following dosing with VMX-C001(UFH cohort) | Up to Day 6
  Change from baseline in thrombin time
Change in prothrombin time (PT) following dosing with VMX-C001 | Up to End of Study (Day 32/33)
  Change from baseline in PT
Change in activated partial thromboplastin time (aPTT) following dosing with VMX-C001 | Up to End of Study (Day 32/33)
  Change from baseline in aPTT
Change in fibrinogen following dosing with VMX-C001 | Up to End of Study (Day 32/33)
  Change from baseline in fibrinogen
Change in dilute Russell viper venom time (dRVVT) following dosing with VMX-C001(UFH Cohort only) | Up to Day 6
  Change from baseline in dRVVT
Change in dilute prothrombin time (dPT) following dosing with VMX-C001 (UFH Cohort only) | Up to Day 6
  Change from baseline in dPT
Change in thrombin generation following dosing with VMX-C001 | Up to Day 6
  Change from baseline in thrombin generation measured by calibrated automated thrombography
Change in real time activated clotting time (ACT) following dosing with VMX-C001 (UFH cohort only) | Up to Day 6
  Change from baseline in ACT
Change in anti-factor 10a (FXa) activity following dosing with VMX-C001 (LMWH Cohort only) | Up to Day 6
  Change from baseline in anti-FXa activity

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No